CLINICAL TRIAL: NCT07023107
Title: Pericapsular Nerve Group Block Mitigates Surgical Stress and Enhances Analgesia in Total Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: NLR and PLR Levels Following PENG Block in Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7/2025
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-06

CONDITIONS: Hip Arthropathy; Hip Osteoarthritis; Hip Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Sodium Chloride; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham blocks (Placebo Comparator): PENG block with 20ml of 0.9% sodium chloride
  Interventions: Drug: 0.9% Sodium Chloride Injection
- PENG block (Active Comparator): PENG block with 20ml 0f 0.2% ropivacaine
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution

INTERVENTIONS:
Drug: 0.9% Sodium Chloride Injection — After spinal anesthesia, the ultrasound-guided PENG block will be performed with 20ml of 0.9% sodium chloride
  Arms: Sham blocks
Drug: Ropivacaine 0.2% Injectable Solution — After spinal anesthesia, the ultrasound-guided PENG block will be performed with 20 ml of 0.2% ropivacaine
  Arms: PENG block

SUMMARY:
Effect of PENG block on NLR and PLR following hip arthroplasty

DETAILED DESCRIPTION:
The NLR is a sensitive indicator of inflammation confirmed in numerous studies and has a predictive and prognostic value. NLR is a cheap, simple, fast-acting, readily available stress and inflammation parameter with high sensitivity and low specificity. Dynamic changes in the NLR precede the clinical state by several hours and may alert clinicians to the ongoing pathological process early. NLR is a new promising marker of cellular immune activation, an important indicator of stress and systemic inflammation. It opens a new dimension for clinical medicine, enabling a better understanding of the biology of inflammation, the linkage and antagonism between innate and adaptive immunity, and their clinical consequences for health and disease.

NLR is affected not only by surgical trauma but also by the method of anesthesia. In recent years, the influence of regional anesthesiology on reducing the inflammatory response after surgical procedures has been emphasized. However, there have been very few studies evaluating the effect of various methods of anesthesia on the NLR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA classification I-III
* Aged 60-100 years
* Who will be scheduled for hip arthroplasty under spinal anesthesia

Exclusion Criteria:

* Patients who have a history of bleeding diathesis
* Take anticoagulant therapy
* History of chronic pain before surgery
* Multiple trauma
* patients unable to assess their pain (dementia)
* patients operated under general anesthesia
* patients having an infection in the region of the procedure
* the patient who does not accept the procedure

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Neutrophil-to-lymphocyte ratio | 12 hours after surgery
  Neutrophil to lymphocyte ratio (NLR) is used as a marker of subclinical inflammation. It is calculated by dividing the number of neutrophils by number of lymphocytes, usually from peripheral blood sample, but sometimes also from cells that infiltrate tissue, such as tumor.

SECONDARY OUTCOMES:
PLR | 12 hours after surgery
  Platelet-to-lymphocyte ratio
PLR | 24 hours after surgery
  Platelet-to-lymphocyte ratio
PLR | 48 hours after surgery
  Platelet-to-lymphocyte ratio
NLR | 24 hours after surgery
  Neutrophil-to-lymphocyte ratio
NLR | 48 hours after surgery
  Neutrophil-to-lymphocyte ratio
first need of opiate | 48 hours after procedure
  Time after surgery when the patient needs opiate for the first time
Opioid Consumption | 48 hours after surgery
  Total opiate consumption after surgery
Pain score | 4 hours after surgery
  NRS (Numerical Rating Scale) - ranging from 0 to 10, where 0 represents "no pain" and 10 represents the "worst pain imaginable"
Pain score | 8 hours after surgery
  NRS (Numerical Rating Scale) - ranging from 0 to 10, where 0 represents "no pain" and 10 represents the "worst pain imaginable"
Pain score | 12 hours after surgery
  NRS (Numerical Rating Scale) - ranging from 0 to 10, where 0 represents "no pain" and 10 represents the "worst pain imaginable"
Pain score | 24 hours after surgery
  NRS (Numerical Rating Scale) - ranging from 0 to 10, where 0 represents "no pain" and 10 represents the "worst pain imaginable"

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, M.D. Ph.D., Study Chair — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes